CLINICAL TRIAL: NCT00073255
Title: Evaluation of Tolerability, Safety, and Pharmacokinetics of hOKT3g1 (Ala-Ala)
Brief Title: Safety and Pharmacokinetics (PK) of hOKT3g1 (Ala-Ala) in Type 1 Diabetes Mellitus (T1DM)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ITNO17AI (completed)
Record Dates: First submitted 2003-11-18; First posted 2003-11-20 (Estimated); Last update posted 2010-01-15 (Estimated); Status verified 2010-01

CONDITIONS: Diabetes Mellitus, Insulin-Dependent
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — alanylalanine

INTERVENTIONS:
Drug: hokt3g1 (ALA-ALA)

SUMMARY:
To assess the tolerability and safety of hOKT3g1 (Ala-Ala) after a 12-day dosing regimen administered via intravenous infusion. To assess the pharmacokinetics of hOKT3g1 (Ala-Ala).

ELIGIBILITY:
To be eligible

* participants will have Type 1 diabetes, diagnosed within the previous 12 months and established by standard American Diabetes Association criteria.
* All participants will have autoantibodies: either anti-GAD65, anti-ICA512, or if treated with insulin for less than 7 days, anti-insulin.
* The age range will be between 8 and 30 years; and
* a minimum weight of 34 kg.

Ages: 8 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 12
Dates: Start 2003-06; Study Completion 2005-12

CONTACTS AND LOCATIONS:
Locations (1):
- Columbia University, New York, New York, United States